CLINICAL TRIAL: NCT06058897
Title: Cerebral MRI Markers and Oculomotor Indices in Human Ageing: Potential Predictors of Cognitive Maintenance or Decline
Brief Title: Magnetic Resonance Imaging (MRI) and Eye-tracking Predictive Markers of Cognitive Ageing.
Acronym: PrediCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0357
Record Dates: First submitted 2023-06-22; First posted 2023-09-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aging
Keywords: ageing; locus coeruleus; noradrenaline; cognition; memory; MRI; pupillometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): MRI, eye-tracking and cognitive exams will be completed by subjects.
  Interventions: Other: MRI; Other: eye-tracking; Other: cognitive exams

INTERVENTIONS:
Other: MRI — MRI examinations will be conducted on the 3T MRI technical platform. During the MRI examination, images reflecting the integrity of the LC (quantification of neuromelanin as well as its functional connections with the different brain regions (resting functional MRI) will be acquired. High-resolution T1 and T2 weighted images of the the entire brain will also be acquired for the volumetry of cerebral areas.
Other: eye-tracking — Eye tracking examinations will be conducted using an EyeBrain medical device (class IIa) developed by Suricog. This eye tracker will be installed in a box, in an experimental room. The eye tracker is combined with a computer to present visual cognitive tasks. Pupillary dilation/constriction measurements will be acquired at rest (when fixing a cross presented on the screen) and during the performance of different cognitive tasks (exploration and processing of scenes visuals, reading texts, making saccades or anti-saccades when presenting visual targets). These pupillary measurements will then be linked to the memorization of the stimuli presented, this recognition being tested at the end of the exam.
Other: cognitive exams — Cognitive measures will be acquired during an evaluation session through interactive cognitive exercises. These exercises are developed using tools offered by Covirtua Healthcare (Covirtua Cognition software). Some exercises will test cognitive systems a priori dependent on NA release (episodic memory, working memory, selective attention, selective inhibition, planning) and other a priori independent of NA (semantic memory: categorization, naming).

SUMMARY:
This research proposes to investigate physiological and cognitive markers of locus coeruleus (LC) neuronal integrity and function in cognitively-healthy participants over 60 years old. The locus coeruleus is a brainstem nucleus, sole source of noradrenaline for the brain. Tau pathology appears in neurons of this nucleus, which may induce initial cognitive changes. The study aims at relating locus coeruleus markers, assessed with MRI and eye-tracking techniques, with cognitive function.

DETAILED DESCRIPTION:
The LC is a small brainstem nucleus, sole source of noradrenaline (NA) to the brain. NA is involved in the physiological arousal response: LC neuronal activity is closely related with pupil dilation, and pupil size is now considered a reliable and easy-access biomarker of LC function. NA-dependent cognitive functions include attention, flexibility and memory, which are selectively impaired with age. Accordingly, LC-NA system dysfunction may occur and contribute to initial cognitive changes during old age.

The study will assess, in cognitively-healthy older volunteers from the INSPIRE cohort (n=100, over 60 years old), MRI and pupillometry markers of LC integrity, LC-forebrain connectivity and LC activity. We aim at investigating the relationship between LC biomarkers and cognitive status. Four experimental visits will be conducted by each participant, every 6 months over an 18-month period. Visits V1 and V4 will include MRI, eye-tracking and detailed cognitive exams. Visits V2 and V3 will include a detailed cognitive exam.

ELIGIBILITY:
Inclusion Criteria:

* INSPIRE cohort participant
* Mini-Mental State Examination score ≥ 27 on 30
* Access to a web connection from participant's or relative's home and regular use of web surfing
* Signature of the informed consent
* Affiliated to a social security scheme

Exclusion Criteria:

* Any contra-indications to MRI exam
* Ophthalmic pathology impacting eye-tracking measures
* Neurological or psychiatric pathology
* Person under guardianship or curatorship

Contraindications to MRI examination:

* Pacemaker or cardiac defibrillator
* Implanted material activated by an electrical, magnetic or mechanical system
* Haemostatic clips for intracerebral aneurysms or carotid arteries
* Orthopedic implants
* Claustrophobia

Ophthalmological pathologies impacting eye tracking measurements:

* Glaucoma
* Age-related macular degeneration
* Unoperated cataract

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2028-03-22 (Estimated); Study Completion 2028-03-22 (Estimated)

PRIMARY OUTCOMES:
Imaging contrast between the LC nucleus and the pontine tegmentum region | 18 months
  The outcome will be measured with brainstem anatomical MRI (no unit) at visits V1 (immediately after inclusion) and V4 (18 months after inclusion).

SECONDARY OUTCOMES:
Z-score of the LC-forebrain connectivity at rest | 18 months
  It will be assessed with resting-state functional MRI (no unit) at visits V1 (immediately after inclusion) and V4 (18 months after inclusion).
Amplitude of the phasic pupil response during completion of cognitive tasks | 18 months
  It will be assessed with eye-tracking (in millimeter) at visits V1 (immediately after inclusion) and V4 (18 months after inclusion).
Latency of saccadic eye movements during completion of cognitive tasks | 18 months
  It will be assessed with eye-tracking (in milliseconds) at visits V1 (immediately after inclusion) and V4 (18 months after inclusion).
Amplitude of saccadic eye movements during completion of cognitive tasks | 18 months
  It will be assessed with eye-tracking (in millimeter) at visits V1 (immediately after inclusion) and V4 (18 months after inclusion).
Composite cognitive (executive and memory) score | 18 months
  It will be assessed (no unit) at visits V1 (immediately after inclusion), V2 (6 months after inclusion), V3 (12 months after inclusion) and V4 (18 months after inclusion).
Levels of blood phospho-Tau | 18 months
  It will be assessed by single-molecule array (Simoa) technology (picogram/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PAYOUX, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France